CLINICAL TRIAL: NCT01460602
Title: Phase 1/2 Study of VELCADE (Bortezomib), Nipent (Pentostatin), and Rituxan (Rituximab) (VNR) in Subjects With Relapsed Follicular, Marginal Zone, and Mantle Cell Lymphoma
Brief Title: Velcade, Nipent, Rituxan (VNR) in Subjects With Relapsed Follicular, Marginal Zone, and Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator has relocated to MD Anderson
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Glenn Mills, Professor of Medicine, Louisiana State University Health Sciences Center Shreveport
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05266
Record Dates: First submitted 2010-06-10; First posted 2011-10-27 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-07

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma
Keywords: Lymphoma; Follicular; Marginal Zone; Mantle Cell; Velcade; bortezomib; Nipent; pentastatin; Rituxan; rituximab; Turturro; Shreveport
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma | interventions — Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: establish MTD (Experimental): Part 1 consists of dosing to determine maximum tolerated dose (MTD) and dose limiting toxicity (DLT).
  Interventions: Drug: MTD of Velcade, Nipent and Rituxan established in Part 1
- Part 2: The MTD from Part 1 (Experimental): During the Phase 2 part of the study, approximately 24 additional subjects will be enrolled in order to obtain a total of 30 response-evaluable subjects treated at the maximum tolerated dose.
  Interventions: Drug: MTD of Velcade, Nipent and Rituxan established in Part 1

INTERVENTIONS:
Drug: MTD of Velcade, Nipent and Rituxan established in Part 1 — One of the following dose levels will be chosen and used in Part 2:
  1. (VAN1) VA= 1.3 mg/m2 IV Days 1, 4, 8, 11 N1= 2 mg/mg2 IV Days 1, 8 375 mg/m2 IV Day 1
  2. (VAN2) VA= 1.3 mg/m2 IV Days 1, 4, 8, 11 N1= 4 mg/mg2 IV Days 1, 8 375 mg/m2 IV Day 1
  3. (VBN1) VA= 1.5 mg/m2 IV Days 1, 4, 8, 11 N1= 2 mg/mg2 IV Days 1, 8 375 mg/m2 IV Day 1
  4. (VBN2) VA= 1.5 mg/m2 IV Days 1, 4, 8, 11 N1= 4 mg/mg2 IV Days 1, 8 375 mg/m2 IV Day 1

SUMMARY:
This is a phase 1/2 Study of VELCADE (bortezomib), Nipent (pentostatin), and Rituxan (rituximab) (VNR) in Subjects with Relapsed Follicular, Marginal Zone, and Mantle Cell Lymphoma.

DETAILED DESCRIPTION:
Number of Subjects: During the Phase 1 part of the study as many as 15 subjects may be enrolled, based on the dose escalation scheme; the actual number of subjects enrolled will depend on the dose level at which the maximum tolerated dose (MTD) is established.

During the Phase 2 part of the study, approximately 15 subjects will be enrolled in order to obtain a total 30 response-evaluable subjects.

Study Objectives:

The primary objectives of this study are:

• Assess the CR and ORR following treatment with VELCADE (bortezomib), Nipent (pentostatin) and Rituxan (rituximab) (VNR) in subjects with follicular lymphoma (FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL) who have relapsed or been refractory after receiving at least 1 prior therapy.

The secondary objectives of this study are to:

* Determine the MTD of VELCADE and Nipent in combination with Rituxan (VNR) in subjects with follicular lymphoma (FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL) who have relapsed or been refractory after receiving at least 1 prior therapy
* Evaluate the safety and tolerability of VNR
* Determine the time to response
* Determine duration of response
* Determine the time to progression (TTP)
* Determine the progression free survival (PFS) rate
* Determine the 1-year survival
* Determine overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent.
2. Male or female subject 18 years of age and older
3. Karnofsky Performance Status (KPS) score of 50%. ECOG Performance Status score greater than 2.
4. Histologically confirmed follicular Grade 1-3a, marginal zone or mantle cell NHL.
5. Relapsed or progressive disease after at least 1 prior chemotherapy requiring treatment.
6. Bi-dimensionally measurable disease with at least 1 lesion 2 cm in a single dimension
7. Hematologic, hepatic, and renal function parameters.
8. Recovered fully from any significant toxicity associated with prior surgery, radiation treatments, chemotherapy, biological therapy, autologous bone marrow or stem cell transplant, or investigational drugs
9. Expected survival of 3 months
10. Accepted birth control methods during treatment and for 12 months after completion of treatment.

Exclusion Criteria:

1. Follicular lymphoma Grade 3b
2. History of allergy to any of the study medications, their analogues, murine proteins, or excipients in the various formulations
3. Grade 2 peripheral neuropathy or clinical examination within 14 days before enrollment
4. Serum creatinine 2.5 mg/dL within 14 days before enrollment.
5. Absolute neutrophil count (ANC) < 1,000/L, platelet count < 70,000/L within 14 days before enrollment
6. Aspartate transaminase (AST [SGOT]) and alanine transaminase (ALT/SGPT]) > 2 x the upper limit of normal (ULN), total bilirubin > 3 ULN
7. Rituxan refractory or refractory to anti-CD20 radioimmunotherapy (no response to prior Rituxan or prior Rituxan-containing regimen, or a response with a TTP of less than 6 months)
8. Cancer radiotherapy, biological therapy, or chemotherapy within 3 weeks prior to Study Day 1 (6 weeks if nitrosurea or mytomycin-C)
9. Prior lymphoma vaccine therapy within 12 months to Study Day 1
10. Prior antibody therapy for lymphoma (including radioimmunotherapy) within 6 months prior to Study Day 1
11. Autologous bone marrow or stem cell transplant within 6 months prior to Study Day 1
12. Known history of hepatitis or hepatic disease.
13. Presence of central nervous system (CNS) lymphoma
14. Known history of HIV infection or AIDS
15. Histologic transformation (Follicular or Marginal zone to diffuse large B cell lymphoma [DLBCL]
16. Presence of pleural or peritoneal effusion with positive cytology for lymphoma
17. Another primary malignancy requiring active treatment
18. Serious non-malignant disease (e.g., congestive heart failure [CHF], hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions (including psychiatric), which would compromise protocol objectives n the opinion of the Investigator and/or Sponsor
19. New York Heart Association Class III or IV (Appendix D) cardiac disease
20. Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1
21. Female subject who is pregnant or currently breast-feeding
22. Received other investigational drugs with 14 days before enrollment
23. Hypersensitivity to bortezomib, pentostatin, rituximab, boron or mannitol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
CR following treatment with VELCADE(bortezomib)/Nipent(pentostatin/Rituxan (rituximab)(VNR) in subjects with follicular lymphoma(FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL)relapsed or refractory after at least 1 prior therapy | up to 48 months
  Study Days 1, 4, 8, 11 of 6 cycles (up to 3 weeks each) and Days 63/126, then Study Months 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48
ORR following treatment with VELCADE(bortezomib)/Nipent(pentostatin/Rituxan (rituximab)(VNR) in subjects with follicular lymphoma(FL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL)relapsed or refractory after at least 1 prior therapy | up to 48 months
  Study Days 1, 4, 8, 11 of 6 cycles (up to 3 weeks each) and Days 63/126, then Study Months 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48

SECONDARY OUTCOMES:
Maximum Tolerated Dose | Study Days 1, 4, 8, 11 of 6 cycles (up to 3 weeks each) and Days 63/126, then Study Months 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48
  Number of participants with adverse events as a measure of safety and tolerability
Rate of progression of disease | Study Days 1, 4, 8, 11 of 6 cycles (up to 3 weeks each) and Days 63/126, then Study Months 6, 9, 12, 15, 18, 21, 24, 30, 36, 42 and 48
  Summary data on time to progression of disease of study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Turturro, MD, Principal Investigator — LSUHSC-S
Locations (1):
- LSU - Shreveport Health Sciences Center, Feist-Weiller Cancer Center, Shreveport, Louisiana, United States